CLINICAL TRIAL: NCT06016192
Title: Medical Rehabilitation of Patients With Long-term Post-Covid-19 Syndrome - a Comparison of Aerobic Interval and Continuous Training
Brief Title: Aerobic Training for Rehabilitation of Patients With Post Covid-19 Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witten/Herdecke (Other)
Collaborators: Institut für Rehabilitationsforschung Norderney (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCS_Training_01
Record Dates: First submitted 2023-08-28; First posted 2023-08-29 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Post-COVID-19 Syndrome; Long-COVID-19 Syndrome
Keywords: COVID-19; Fatigue; Rehabilitation; Exercise Training; Infectious Disease
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Fatigue; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Two-arm randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous aerobic training (Active Comparator): Moderate continous endurance training, ergometer
  Interventions: Behavioral: Aerobic Exercise Training
- Interval aerobic training (Experimental): Moderate intensity interval training, ergometer
  Interventions: Behavioral: Aerobic Exercise Training

INTERVENTIONS:
Behavioral: Aerobic Exercise Training — Physical activity performed as controlled aerobic exercise training on ergometer

SUMMARY:
Post-COVID-19 syndrome (PCS) occurs as a sequelae after acute infection with the SARS-CoV-2 virus (COVID-19 infection). PCS is defined as symptom persistence over a period of 12 weeks from infection and/or the appearance of new symptoms in this period. While the majority of affected patients experience a gradual healing process without targeted treatment, the need for effective medical rehabilitation is high at least for patients with persistent PCS.

Given that physical exercise has been shown to be beneficial in multiple pathologies such as cardiovascular diseases, neuropathic disorders, and pulmonary diseases it has been suggested that physical exercise including aerobic training could exert beneficial effects also in PCS. This study aims to analyse the use of moderate-intensity aerobic exercise training for medical rehabilitation of PCS patients.

DETAILED DESCRIPTION:
Post-COVID-19 syndrome (PCS) is a condition that occurs following an acute infection with the SARS-CoV-2 virus (COVID-19). PCS is characterized by symptom persistence for at least 12 weeks after the infection or the emergence of new symptoms during this period. Current guidelines propose several criteria for diagnosing PCS, including persistent symptoms from the acute COVID-19 phase, new symptoms leading to health limitations, symptoms assumed to be related to COVID-19 after the acute phase, and worsening of pre-existing underlying conditions. PCS is a complex and multisystemic disorder, with symptoms ranging from chronic fatigue, decreased physical performance, muscular weakness, and pain to cognitive impairment (often referred to as brain fog) and mental and psychological distress resembling a post-traumatic stress reaction. The exact causes of PCS are not fully understood but may involve processes such as endothelial dysfunction, cytokine storm, and increased oxidative stress affecting various organs and structures in the body. The incidence of PCS varies depending on the population studied and the severity of symptoms considered, with estimates ranging from 7.5% to 41% among non-hospitalized patients with acute infection.

Medical rehabilitation is essential for patients with persistent PCS, but there are limited studies on its efficacy, especially in the context of aerobic endurance training. Physical exercise, including aerobic training, has shown positive effects in various diseases, and it is suggested that it may be beneficial for PCS as well. However, there is limited evidence regarding the effectiveness of aerobic endurance training in reducing the burden of decreased physical performance in PCS. Moreover, there is a lack of guidelines for PCS patients related to exercise-based rehabilitation. Aerobic endurance training has been proven to have positive effects on multiple physiological functions and is recommended for chronic heart and pulmonary diseases. Studies have also suggested that aerobic interval training may be advantageous for PCS patients, as it reduces ventilatory demand and may alleviate dyspnea and breathing effort. This study aims to investigate the efficacy of moderate-intensity aerobic endurance training performed as either continuous training and interval training for the medical rehabilitation of PCS patients.

The study will include PCS patients referred for inpatient medical rehabilitation in Germany with a history of (at least one) Covid-19 infection and ongoing or newly expressed performance deficits lasting for at least 3 months prior to recruitment. Performance deficits will be documented according to the recent consensus statement, with the cluster of lead symptoms including fatigue/exercise intolerance, shortness of breath, and cognitive dysfunction impairing activity of daily living and everyday functioning. A detailed clinical workup will be performed, and the history of comorbidities and current medication will be documented. After admission, patients will be randomized to a continuous training (CT) or interval training (IT) group. Patients will receive individual medical rehabilitation including a combination of strength, respiratory and cognitive training, as well as physio-, psycho- and nutrition therapy, unaltered for both groups. Data on medical rehabilitation including prescriptions of therapeutic actions and participation will be recorded for all patients. Symptom-limited spiroergometry at admission and after 4-6 weeks of inpatient rehabilitation (before discharge) will be performed to analyze improvements in exercise capacity. Validated questionnaires will be used to document patients' disease perception.

ELIGIBILITY:
Inclusion Criteria:

* a history of (at least one) Covid-19 infection
* ongoing or newly expressed performance deficits lasting for at least 3 months prior to recruitment
* referral to inpatient rehabilitation
* signed informed consent

Exclusion Criteria:

* unstable condition
* incapable of understanding study information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Cardiorespiratory Fitness (CRF) | Baseline and week 4 (i. e. before discharge)
  CRF will be measured as peak oxygen uptake (VO2peak) determined by spiroergometry

SECONDARY OUTCOMES:
Change in Submaximal Cardiorespiratory Fitness (CRF) | Baseline and week 4 (i. e. before discharge)
  Submaximal CRF will be measured as submaximal oxygen uptake (VO2 at ventilatory threshold 1 [VT1]) determined by spiroergometry
Change in Fatigue | Baseline and week 4 (i. e. before discharge)
  Fatigue will be assessed using the "The Multidimensional Fatigue Inventory (MFI20)".
Work requirements and workload | Baseline
  Work requirements and workload will be assessed using the "Workability Index (WAI)".
Change Health-related quality of life | Baseline and week 4 (i. e. before discharge)
  Health-related quality of life will be assessed using the "RAND 36-Item Health Survey (SF-36)".
Wellbeing | Baseline and week 4 (i. e. before discharge)
  Wellbeing will be assessed using the "WHO-5 Well-Being Index".
Change in Depression and Anxiety | Baseline and week 4 (i. e. before discharge)
  Depression and Anxiety will be assessed using the Hospital Anxiety and Depression Scale (HADS)

OTHER OUTCOMES:
Change in training load | Daily, from baseline to week 4 (i. e. before discharge)
  Training load will be assessed by analysis of documented ergometer settings (mean Watts)
Training participation | Daily, from baseline to week 4 (i. e. before discharge)
  Training participation will be assessed by number of performed ergometer training sessions
Change in minute ventilation (VE) | Baseline and week 4 (i. e. before discharge)
  Minute ventilation will be determined by spiroergometry measuring breath-by-breath volumes (ml)
Change in carbon dioxide production (VCO2) | Baseline and week 4 (i. e. before discharge)
  Carbon dioxide production (VCO2) will be determined by spiroergometry measuring breath-by-breath volumes of exhaled carbon dioxide (ml)
Change in submaximal and maximal workload (Watt) | Baseline and week 4 (i. e. before discharge)
  Submaxmal and maximal workload (Watt) will be determined by spiroergometry

CONTACTS AND LOCATIONS:
Locations (1):
- Clinic Königsfeld, Ennepetal, North Rhine-Westphalia, Germany